CLINICAL TRIAL: NCT02773485
Title: Phase III Randomized Trial of High Dose Chemoradiation and Systemic Chemotherapy vs Systemic Chemotherapy Alone in Patients With Unresectable Nonmetastatic Cholangiocarcinoma
Brief Title: Chemo Alone or in Combination With Radiation in Unresectable Cholangiocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Associate Professor, Radiation Oncology, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC IRB 1457
Record Dates: First submitted 2016-03-08; First posted 2016-05-16 (Estimated); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Radiation; Neoadjuvant Therapy; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Systemic Chemotherapy (Active Comparator): Irrespective of arm allocation Baseline Positron Emission Tomography(PET) scan and hepatic function assessment will be done. Those randomized to this arm will receive systemic chemotherapy delivered on day 1 and 8 every 3 weekly, with gemcitabine 1000 mg/m2 and cisplatin 25 mg/m2. After first 4 cycles patients will undergo repeat Contrast Enhanced Computed Tomography(CECT)/PET scan. If CECT/PET scan shows stable/ responding disease then patients will continue to receive the same chemotherapy. In case of locally progressive/ systemic disease on chemotherapy patients may be considered for second line palliative chemotherapy or best supportive care. The use of radical chemoradiation is not allowed on disease progression in this arm. However palliative radiation may be used.
  Interventions: Drug: Systemic chemotherapy
- Chemotherapy and radiation (Experimental): In those randomized to radiation arm with receive high dose radiation with Intensity Modulated Radiation Therapy in addition to systemic and concurrent chemotherapy. The gross tumor will comprise the high dose volume. The adjacent areas of suspected microscopic disease will form the low dose volume. When only external radiation is used the aim will be to deliver 52.5-60 Gy/ 25 fractions to the gross disease and 45 Gy/ 25 fractions to suspected microscopic disease along with weekly gemcitabine (300 mg/ m2) .
  Interventions: Radiation: High Dose Radiation; Drug: Systemic chemotherapy

INTERVENTIONS:
Radiation: High Dose Radiation — The aim will be to deliver 52.5-60 Gy/ 25 fractions to the gross disease and 45 Gy/ 25 fractions to suspected microscopic disease along with weekly gemcitabine (300 mg/ m2) .
  Other Names: Radiation
  Arms: Chemotherapy and radiation
Drug: Systemic chemotherapy — This arm will receive maximum 8 cycles of gemcitabine 1000 mg/m2 and cisplatin 25 mg/m2 delivered on day 1 and 8 every 3 weekly.
  Other Names: Gemcitabine and Cisplatin regimen

SUMMARY:
The study evaluates impact of high dose radiation on overall survival in patients with unresectable nonmetastatic cholangiocarcinoma. The study randomizes patient between systemic chemotherapy alone and systemic chemotherapy and high dose radiation

DETAILED DESCRIPTION:
Currently the standard of care of unresectable non-metastatic cholangiocarcinoma is chemotherapy which has a median survival of 11.7 months (ABC-02 study). While this study included almost 60% of patients with cholangiocarcinomas (intrahepatic, extra hepatic and hilar), almost 73-76% of patients in each arm had metastases to begin with. And while the overall survival of the entire cohort was significantly improved by gemcitabine plus cisplatin compared to cisplatin alone, the hazard ratios for intrahepatic {0.57 (0.34-0.94)}, extra hepatic {0.73 (0.43-1.23)} and hilar cholangiocarcinomas {0.59 (0.32-1.09)} were all insignificant. Even though concurrent chemoradiation+/= brachytherapy has been used for management of cholangiocarcinomas for more than 3 decades the lack of level I evidence prevents from it being recommended as the first line management across multidisciplinary clinics.

While either modality alone rarely yields survival of more than 12 months, recent reports of improved median survival with combination of high dose radiation and systemic chemotherapy necessitates investigation into role of combination of high dose (chemo) radiation and systemic chemotherapy.

All patients with diagnosis of nonmetastatic unresectable cholangiocarcinoma who fulfill the study eligibility criteria will be evaluated for study participation. Patients will undergo upfront randomization into one of the study arms (systemic chemotherapy alone vs Systemic chemotherapy+ High dose radiation) The study stratification criteria will be done according the primary site i.e. Intrahepatic vs Extrahepatic.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Performance Status 0-2
* Tissue diagnosis of adenocarcinoma of the biliary tract. Wherever tissue diagnosis is not feasible in spite of repeated attempts a multidisciplinary consensus on clinicoradiological diagnosis of cholangiocarcinoma (CA 19-9= 100mg/ml with a radiological evidence of malignant stricture) should be made and patients consent should be available for treatment without tissue diagnosis.
* Unresectable disease as determined by hepatobiliary surgical team.
* No evidence of peritoneal or distant metastasis.
* No radiological evidence of paraaortic nodal disease.
* Child A or Child B (score 7)
* Ability to tolerate radical treatment.

Exclusion Criteria:

* Multicentric intrahepatic cholangiocarcinoma (however adjacent satellite lesions are permitted)
* Inability to deliver safe radiation due to high tumor/ liver ratio.
* Active cholangitis.
* Expected Survival<6 months.
* Unresolved biliary tract obstruction.
* Inability in deliver systemic chemotherapy (persistent bilirubin>3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2015-05; Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 years from completion of study
  The trial is designed to assess a 36 month benefit overall survival

SECONDARY OUTCOMES:
loco-regional progression free survival | 3 years from completion of accrual
  Will compare the loco-regional progression free survival between both the arms
Toxicity Assessment | upto 3 years
  Assessment will be done according to CTCAE v4.0
Quality of Life Assessment of patients over a period of time | 3 years from completion of accrual
  Assessment will be done according to Fact-Hep(version 4)
Surgical Resectability Rates | 6 weeks from completion of primary treatment
  To assess the number of patient who can be taken for surgery in view of good response after treatment
cause specific survival | 3 years from completion of accrual
  Will compare the cause specific survival between both the arms

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Chopra, MD, Principal Investigator — ACTREC,Tata Memorial Centre
Locations (1):
- Advanced Centre of Treatment Research and Education In Cancer,Tata Memorial Centre, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided